CLINICAL TRIAL: NCT03911232
Title: The Improvement of Intraoperative Neuromonitoring of Recurrent Laryngeal Nerve During Thyroid Surgery
Brief Title: The Improvement of Intraoperative Neuromonitoring of Recurrent Laryngeal Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, I-Cheng Lu, Doctor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KMUH-IRB-E-20150023
Record Dates: First submitted 2016-12-05; First posted 2019-04-11 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Intra-Operative Injury
Keywords: intraoperative neural monitoring
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Enhanced recovery (Experimental): rocuronium 2 effective dose at anesthesia induction sugammadex after skin incision and before extubation (total 2 mg/kg iv)
  Interventions: Drug: sugammadex
- Conventional anesthesia (No Intervention): standard general anesthesia protocol (1 effective dose of rocuronium at anesthesia induction)

INTERVENTIONS:
Drug: sugammadex — standard general anesthesia protocol with sugammadex
  Other Names: Bridion
  Arms: Enhanced recovery

SUMMARY:
Objectives: The use of neuromuscular blocking agent may interfere with the function of intraoperative neuromonitoring (IONM) in thyroid surgery.

DETAILED DESCRIPTION:
An enhanced neuromuscular-blockade (NMB) recovery protocol was investigated in a clinically applied during thyroid neural monitoring surgery. In as subsequent clinical application study, 60 patients who underwent thyroidectomy with IONM followed an enhanced NMB recovery protocol- rocuronium 0.6 mg/kg at anesthesia induction and sugammadex 2 mg/kg at operation start. Train-of-four (TOF) ratio was used for continuous quantitative monitoring of neuromuscular transmission.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing intraoperative neuromonitoring of recurrent laryngeal nerve during thyroidectomy

Exclusion Criteria:

* Patients with a history of significant cardiac, pulmonary, hepatic, or renal disease, body mass index <18.5 or >35, chronic drug or alcohol abuse

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
sugammadex 2 mg/kg allows effective and rapid restoration of neuromuscular function suppressed by rocuronium | 1 month each case
  Electromyography signal to assess the quality of neuromonitoring

CONTACTS AND LOCATIONS:
Locations (1):
- I-Cheng Lu, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No